CLINICAL TRIAL: NCT06673654
Title: A Multi-Center, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Study, Comparing Ruxolitinib Topical Cream 1.5% (Taro Pharmaceuticals U.S.A, Inc.) to OPZELURA (Ruxolitinib) Cream and Both Active Treatments to a Placebo Control in the Treatment of Mild-to-Moderate Atopic Dermatitis.
Brief Title: A Study, Comparing Ruxolitinib Topical Cream 1.5% (Taro Pharmaceuticals U.S.A, Inc.) to OPZELURA (Ruxolitinib) Cream for the Treatment of Mild-to-Moderate Atopic Dermatitis.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RXLC-2118
Record Dates: First submitted 2024-11-02; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2023-10

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — ruxolitinib

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Ruxolitinib Topical Cream 1.5% (Experimental): The investigational product is to be self-administered by applying a thin layer twice daily to cover the affected areas up to 20% body surface area for approximately 8 weeks. The maximum weekly dose of the study drug should not exceed 60 g.
  Interventions: Drug: Ruxolitinib Topical Cream 1.5%
- OPZELURA (Ruxolitinib) Cream (Active Comparator): The investigational product is to be self-administered by applying a thin layer twice daily to cover the affected areas up to 20% body surface area for approximately 8 weeks. The maximum weekly dose of the study drug should not exceed 60 g.
  Interventions: Drug: OPZELURA (Ruxolitinib) Cream
- Placebo Control (Placebo Comparator): The investigational product is to be self-administered by applying a thin layer twice daily to cover the affected areas up to 20% body surface area for approximately 8 weeks. The maximum weekly dose of the study drug should not exceed 60 g.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ruxolitinib Topical Cream 1.5% — The investigational product is to be self-administered by applying a thin layer twice daily to cover the affected areas up to 20% body surface area for approximately 8 weeks. The maximum weekly dose of the study drug should not exceed 60 g.
  Other Names: Test Product
  Arms: Ruxolitinib Topical Cream 1.5%
Drug: OPZELURA (Ruxolitinib) Cream — The investigational product is to be self-administered by applying a thin layer twice daily to cover the affected areas up to 20% body surface area for approximately 8 weeks. The maximum weekly dose of the study drug should not exceed 60 g.
  Other Names: Reference Product
  Arms: OPZELURA (Ruxolitinib) Cream
Drug: Placebo — The investigational product is to be self-administered by applying a thin layer twice daily to cover the affected areas up to 20% body surface area for approximately 8 weeks. The maximum weekly dose of the study drug should not exceed 60 g.
  Other Names: Vehicle
  Arms: Placebo Control

SUMMARY:
To demonstrate the therapeutic equivalence and safety of Ruxolitinib Topical Cream 1.5% (Taro Pharmaceuticals U.S.A, Inc.) and OPZELURA (Ruxolitinib) Cream in the treatment of mild-to-moderate atopic dermatitis

DETAILED DESCRIPTION:
A multi-center, double-blind, randomized, placebo-controlled, parallel-group study, comparing Ruxolitinib Topical Cream 1.5% (Taro Pharmaceuticals U.S.A, Inc.) to OPZELURA (Ruxolitinib) Cream and both active treatments to a placebo control in the treatment of mild-to-moderate atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female aged ≥ 12 years
* Subjects who are 18 years of age or older must have provided IRB approved written informed consent. Subjects 12 to 17 years of age, inclusive, must have provided IRB approved written assent; this written assent must be accompanied by an IRB approved written informed consent from the Subject's legally acceptable representative (i.e., parent or guardian).
* Subjects who have a clinical diagnosis of AD as defined by the criteria of Hanifin and Rajka.
* Subjects who have a clinical diagnosis of AD for at least 2 years.
* Subjects who have IGA Score of 2 (Mild) or 3 (Moderate) for AD severity.
* Subjects who have AD involvement of 3-20% of the body surface area (BSA) and does not include the scalp.

Exclusion Criteria:

* Female Subjects who are pregnant, nursing or planning to become pregnant during study participation.
* Subjects with a history of hypersensitivity or allergy to Ruxolitinib and/or any of the study medication ingredients
* Subjects with unstable course of AD (spontaneously improving or rapidly deteriorating) as determined by the investigator in the 4 weeks prior to baseline.
* Subjects with the presence of any skin condition that would interfere with the diagnosis or assessment of AD (e.g., other types of eczema, pigmentation, or extensive scarring).

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 476 (Actual)
Dates: Start 2023-08-11 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
Demonstration of therapeutic equivalence, superiority, and safety of the Investigational Products. | Baseline to Week 8
  The percentage of subjects in each treatment group with "Treatment Success" (defined as an IGA score of 0 (clear) or 1 (almost clear) with at least a two-point improvement from baseline, at the Week 8 (Day 56 ± 4 days) visit.

CONTACTS AND LOCATIONS:
Overall Officials: Andy Silverman, Study Chair — Catawba Research, LLC
Locations (1):
- Taro Pharmaceuticals USA Inc., Hawthorne, New York, United States

IPD SHARING:
Plan to Share IPD: No